CLINICAL TRIAL: NCT00001038
Title: A Randomized, Double-Blind Trial of Valacyclovir Hydrochloride (BW 256U87) Prophylaxis for Opportunistic Cytomegalovirus End-Organ Disease in Patients With Advanced HIV Infection (< 100 CD4+ Lymphocytes)
Brief Title: A Study of Valacyclovir Hydrochloride in the Prevention of Life-Threatening Cytomegalovirus Disease in HIV-Infected Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Glaxo Wellcome (Industry)
Purpose: Treatment
Other Study IDs: ACTG 204; FDA 104C
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-03-01 (Estimated); Status verified 2011-02

CONDITIONS: Cytomegalovirus Infections; HIV Infections
Keywords: Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome; Antiviral Agents
MeSH Terms: conditions — Cytomegalovirus Infections; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Valacyclovir; Acyclovir

INTERVENTIONS:
Drug: Valacyclovir hydrochloride
Drug: Acyclovir

SUMMARY:
PRIMARY: To evaluate the efficacy of valacyclovir hydrochloride (BW 256U87) in the prevention of cytomegalovirus (CMV) end-organ disease in HIV/CMV co-infected patients with CD4+ lymphocytes < 100 cells/mm3. To assess the impact of BW 256U87, high-dose oral acyclovir and low-dose oral acyclovir on survival.

SECONDARY: To evaluate the effect of BW 256U87 on quality of life, the safety of the drug administered concurrently with standard antiretroviral agents and other essential therapies for the treatment and prevention of opportunistic diseases, and the efficacy of BW 256U87 in suppressing activation of other herpesviruses. To evaluate serologic and virologic risk factors for the development of CMV disease, including assessment of HIV activation, and the risk of developing drug-resistant CMV, HSV, and VZV.

Gastrointestinal absorption of acyclovir is not high enough to prevent CMV disease in patients with advanced HIV disease, although there is evidence that high doses of the drug may extend survival. Valacyclovir, a prodrug that is rapidly converted to acyclovir after oral administration, has a higher absorption rate and may therefore provide inhibitory activity against CMV.

DETAILED DESCRIPTION:
Gastrointestinal absorption of acyclovir is not high enough to prevent CMV disease in patients with advanced HIV disease, although there is evidence that high doses of the drug may extend survival. Valacyclovir, a prodrug that is rapidly converted to acyclovir after oral administration, has a higher absorption rate and may therefore provide inhibitory activity against CMV.

Patients are randomized to receive BW 256U87 alone or acyclovir alone as control at either high-dose or low-dose. The acyclovir controls will provide suppressive therapy for herpes simplex infections and may affect survival.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Recommended:

* PCP prophylaxis.

Allowed:

* Any antiretroviral therapies available by prescription or through expanded access or Treatment IND programs, including combination or sequential use.
* Chemotherapy for Kaposi's sarcoma, lymphoma, or other malignancies IF patient is hematologically stable for at least 30 days prior to study entry.
* Discrete courses of oral or parenteral acyclovir for VZV or HSV infection, not to exceed 21 days per episode (may co-enroll on ACTG 169). For recurrent episodes, open-label acyclovir for a total of 60 days over a 12-month period is allowed. Study drug is interrupted.
* Supportive therapies available by prescription, expanded access, or Treatment IND programs, such as G-CSF, GM-CSF, and erythropoietin.
* Other medications necessary for the patient's welfare, at the discretion of the investigator.

Patients must have:

* HIV infection or AIDS-defining conditions.
* CD4+ count < 100 cells/mm3.
* IgG antibodies to CMV.
* No active CMV disease or history of CMV end-organ disease.
* Consent of parent or guardian if less than 18 years of age.
* Ability to comply with protocol.

NOTE:

* Patients may be co-enrolled in ACTG primary infection Phase II/III studies, ACTG opportunistic infection protocols, or treatment protocols or similar studies sponsored by other research networks as long as those studies do not violate the restrictions placed on concomitant therapies and toxicity management.

Prior Medication:

Allowed:

* PCP prophylaxis.
* Any antiretroviral therapies available by prescription or through expanded access or Treatment IND programs, including combination or sequential use.
* Chemotherapy for Kaposi's sarcoma, lymphoma, or other malignancies.
* Acyclovir.
* Supportive therapies available by prescription, expanded access, or Treatment IND programs, such as G-CSF, GM-CSF, and erythropoietin.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Nausea or vomiting that precludes oral dosing.
* Ocular media opacities that preclude adequate visualization of fundi.
* Pregnancy.
* Known hypersensitivity to acyclovir.
* Known lactose intolerance.

Concurrent Medication:

Excluded:

* Systemic interferons and immunomodulators (including CMV hyperimmune serum/globulin and chronic corticosteroids at doses in excess of physiologic replacement).
* Probenecid.
* Investigational or marketed agents with potential activity against CMV, herpes simplex, and/or Varicella zoster, EXCEPT as specifically allowed.

Patients with the following prior condition are excluded:

* Pre-existing necrotizing retinopathy that may interfere with a subsequent diagnosis of CMV retinitis.

Prior Medication:

Excluded:

* Prior ganciclovir, foscarnet, or any investigational anti-CMV agent including use of foscarnet for acyclovir-resistant herpes.
* Interferons, immunomodulators (other than colony stimulating factors), or CMV hyperimmune globulin within 30 days prior to study entry.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1200
Dates: Primary Completion 1996-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Feinberg J, Study Chair
Locations (35):
- United States (21):
  - Birmingham Veterans Administration Med Ctr, Birmingham, Alabama
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - CARE Ctr / UCLA Med Ctr, Los Angeles, California
  - Highland Gen Hosp / San Francisco Gen Hosp, Oakland, California
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - Kaiser Permanente Med Ctr, San Francisco, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Yale Univ, New Haven, Connecticut
  - Northwestern Univ Med School, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Harvard (Massachusetts Gen Hosp), Boston, Massachusetts
  - Boston Med Ctr, Boston, Massachusetts
  - Washington Univ, St Louis, Missouri
  - Mount Sinai Med Ctr, New York, New York
  - North Central Bronx Hosp / Bronx Municipal Hosp, The Bronx, New York
  - Univ of North Carolina School of Medicine, Chapel Hill, North Carolina
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Girard Med Ctr, Philadelphia, Pennsylvania
  - Univ TX Galveston Med Branch, Galveston, Texas
  - Univ of Washington / Madison Clinic, Seattle, Washington
- Saint Vincent's Hosp Med Centre, Sydney, Australia
- Canada (5):
  - Southern Alberta HIV Clinic / Foothills Hosp, Calgary, Alberta
  - Sunnybrook Health Science Ctr, Toronto, Ontario
  - Toronto Hosp, Toronto, Ontario
  - Montreal Chest Institute, Montreal, Quebec
  - Montreal Gen Hosp, Montreal, Quebec
- Hvidovre Univ Hosp, Hvidore, Denmark
- Services des Maladies Infectieuses, Paris, France
- Universitatsklinikum Rudolf Virchow, Berlin, Germany
- Universita Cattolica del Sacro Cuore, Rome, Italy
- South Hosp, Stockholm, Sweden
- Medizinische Universibatspoliklinik Infekbiologie, Bern, Switzerland
- United Kingdom (2):
  - Royal Free Hosp, London
  - Westminster Hosp, London

REFERENCES:
- [Background] Feinberg JE, Hurwitz S, Cooper D, Sattler FR, MacGregor RR, Powderly W, Holland GN, Griffiths PD, Pollard RB, Youle M, Gill MJ, Holland FJ, Power ME, Owens S, Coakley D, Fry J, Jacobson MA. A randomized, double-blind trial of valaciclovir prophylaxis for cytomegalovirus disease in patients with advanced human immunodeficiency virus infection. AIDS Clinical Trials Group Protocol 204/Glaxo Wellcome 123-014 International CMV Prophylaxis Study Group. J Infect Dis. 1998 Jan;177(1):48-56. doi: 10.1086/513804. PMID 9419169
- [Background] Fry J, Coakley D, Power M, Feinberg J. International collaborative clinical trials: the ACTG 204 experience. Int Conf AIDS. 1996 Jul 7-12;11(2):276 (abstract no ThB4146)
- [Background] Griffiths PD, Feinberg J. Detection of cytomegalovirus in samples from patients enrolled in ACTG 204 / Glaxo Wellcome 123-014. Conf Retroviruses Opportunistic Infect. 1996 Jan 28-Feb 1;3rd:54
- [Background] Brosgart C, Fisher E, Pulling C, Chaloner K, Cohn D, Elsadr W, Verheggen R, Schmetter B, Alston B. Prevalence of asymptomatic CMV retinitis (CMVR) in AIDS patients. Conf Retroviruses Opportunistic Infect. 1999 Jan 31-Feb 4;6th:152 (abstract no 453)
- [Background] Fisher E, Brosgart C, Cohn D, Chaloner K, Pulling C, Alston B, Schmetter B, El-Sadr W. Placebo (PLC)-controlled, multicenter trial of adefovir dipivoxil (ADV) in patients (pt) with HIV disease. . Conf Retroviruses Opportunistic Infect. 1999 Jan 31-Feb 4;6th:160 (abstract no 491)
- [Background] Feinberg JE, Bell WR, Chulay JD. A thrombotic microangiopathy (TMA)-like syndrome in patients with advanced HIV disease in a cytomegalovirus (CMV) prophylaxis trial (ACTG 204). Conf Retroviruses Opportunistic Infect. 1997 Jan 22-26;4th:196 (abstract no 715)
- [Background] Sprenger HG, Law G, Pastoor G, Postma S, Schirm J, Weits J, The TH. Cytomegalovirus antigenemia (CMVAg) compared with other CMV tests during phase III study of valaciclovir (VACV) for CMV prophylaxis in advanced HIV disease (ACTG 204 study). Int Conf AIDS. 1996 Jul 7-12;11(2):285 (abstract no ThB4200)
- [Background] Bell WR, Chulay JD, Feinberg JE. Manifestations resembling thrombotic microangiopathy in patients with advanced human immunodeficiency virus (HIV) disease in a cytomegalovirus prophylaxis trial (ACTG 204). Medicine (Baltimore). 1997 Sep;76(5):369-80. doi: 10.1097/00005792-199709000-00004. No abstract available. PMID 9352739
- [Background] Emery V, Sabin C, Feinberg J, Grywacz M, Knight S, Griffiths P. Quantitative effects of valaciclovir on the replication of cytomegalovirus in patients with advanced HIV disease. Conf Retroviruses Opportunistic Infect. 1999 Jan 31-Feb 4;6th:153 (abstract no 459)
- [Background] Weinberg A, Schneider SA, Clark JC. Acyclovir (ACV) and valacyclovir (VAL) prophylaxis of AIDS patients does not alter cytomegalovirus (CMV) susceptibility to ganciclovir (GCV) or foscarnet (FOS). Program Abstr Intersci Conf Antimicrob Agents Chemother. 1996 Sep 15-18:202 (abstract no I87)
- [Background] Nokta MA, Holland F, De Gruttola V, Emery VC, Jacobson MA, Griffiths P, Pollard RB, Feinberg JE; AIDS Clinical Trials Group, Protocol 204/GlaxoWellcome 123-014, International CMV Prophylaxis Study Group. Cytomegalovirus (CMV) polymerase chain reaction profiles in individuals with advanced human immunodeficiency virus infection: relationship to CMV disease. J Infect Dis. 2002 Jun 15;185(12):1717-22. doi: 10.1086/340651. Epub 2002 May 31. PMID 12085316